CLINICAL TRIAL: NCT00519831
Title: Phase II Study of Vinflunine and Cetuximab in the Second Line Treatment of Stage IIIB/IV Non-Small Cell Lung Cancer
Brief Title: Ph II of Vinflunine and Cetuximab in Second Line Treatment of NSCLC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Drug unavailable
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UNC LCCC 0503; NCT00330031 (obsolete NCT alias)
Record Dates: First submitted 2007-08-21; First posted 2007-08-23 (Estimated); Results first posted 2017-06-09 (Actual); Last update posted 2017-06-09 (Actual); Status verified 2017-05

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Cetuximab; vinflunine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vinflunine + Cetuximab (Experimental): Patients may receive more than 4 cycles of therapy if they continue to demonstrate response to therapy, have limited toxicity, and if the treating physician determines that they are deriving clinical benefit from the treatment. The decision of continuing therapy beyond 4 cycles must be discussed with the principal investigator.
  Interventions: Biological: cetuximab; Drug: vinflunine

INTERVENTIONS:
Biological: cetuximab — 400 mg/m² week 1,then 250 mg/m² weekly
  Other Names: erbitux
Drug: vinflunine — Vinflunine 320 mg/m² every 21 days
  Other Names: Javlor

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as vinflunine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some find tumor cells and help kill them or carry tumor-killing substances to them. Others interfere with the ability of tumor cells to grow and spread. Giving vinflunine together with cetuximab may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving vinflunine together with cetuximab works as second-line therapy in treating patients with stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Estimate the objective response rate in patients receiving vinflunine and cetuximab as second-line therapy for stage IIIB or IV non-small cell lung cancer.

Secondary

* Determine the progression-free survival of patients treated with this regimen.
* Determine the safety of this regimen in these patients.
* Determine the overall survival of patients treated with this regimen.
* Determine the duration of overall response in these patients.

OUTLINE: This is a multicenter study.

Patients receive vinflunine IV over 15-20 minutes on day 1 and cetuximab IV over 60-120 minutes on days 1, 8, and 15. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients with responding disease may receive additional courses beyond 4 courses at the discretion of the principal investigator.

After completion of study therapy, patients are followed periodically for 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC) meeting 1 of the following criteria:

  * Unresectable stage IIIB disease with pleural effusion or pericardial effusion
  * Stage IIIB disease that was treated with chemotherapy alone as first-line therapy
  * Stage IV disease
* Must have documented progression of disease after receiving one cytotoxic chemotherapy regimen for metastatic disease
* At least one lesion that is bidimensionally measurable by CT scan or MRI

  * Must have evaluable disease outside the radiation field

    * New lesions that develop within the radiation field are allowed
* Measurable disease status as defined by RECIST criteria
* Brain metastases allowed provided they have been previously treated and are controlled

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Absolute neutrophil count (ANC) > 1,000/mm³
* Hemoglobin > 8.0 g/dL
* Platelet count > 75,000/mm³
* Creatinine < 2.0 times upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 5 times ULN
* Total bilirubin < 2.5 times ULN
* Prior malignancy allowed provided the patient's life expectancy is best defined by the diagnosis of NSCLC
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for up to 4 weeks after completion of study therapy

Exclusion criteria:

* Peripheral neuropathy ≥ 2
* Severe allergic reaction to prior vinca alkaloid treatment
* Active or uncontrolled infection
* Significant history of uncontrolled cardiac disease, including any of the following:

  * Uncontrolled hypertension
  * Unstable angina
  * Myocardial infarction within the past 6 months
  * Uncontrolled congestive heart failure
  * Cardiomyopathy with decreased ejection fraction
* Severe reaction to prior monoclonal antibody therapy

PRIOR CONCURRENT THERAPY:

Inclusion criteria:

* See Disease Characteristics
* Prior oral tyrosine kinase inhibitor therapy (e.g. gefitinib or erlotinib) allowed

  * Not considered cytotoxic therapy for study eligibility purposes if given alone as first-line therapy
* At least 1 week since prior radiotherapy
* At least 21 days since prior and no other concurrent chemotherapy
* Prior adjuvant therapy allowed provided patient received one cytotoxic chemotherapy regimen as treatment for metastatic disease
* Prior bevacizumab allowed

Exclusion criteria:

* Two or more cytotoxic chemotherapy regimens as treatment for metastatic disease
* Prior therapy with monoclonal antibody directed at the epidermal growth factor receptor (EGFR) pathway
* Prior therapy with a vinca alkaloid in the metastatic setting
* Concurrent bevacizumab
* Other concurrent investigational agent(s)
* Concurrent colony-stimulating factors as primary prophylaxis for the prevention of febrile neutropenia
* Concurrent CYP3A4 inhibitor(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-08; Primary Completion 2008-02 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E. Stinchcombe, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Alamance Oncology/Hematology Associates, LLP, Burlington, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 18 patients were enrolled, 2 patients were consented but not enrolled. 1 patient withdrew and 1 patient was taken off the study due to decline in performance status.
Period: Overall Study
Arm/Group | Vinflunine + Cetuximab
Started | 16
Completed | 13
Not Completed | 3
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Arm/Group | Vinflunine + Cetuximab
Number analyzed (Participants) | 16
Age, Continuous [Median (Full Range); unit: years] | 60.5 [50 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16
Number of Participants who had a score of 0-1 in the The Eastern Cooperative Oncology Group (ECOG) [Count of Participants; unit: Participants] — Measure Description: A scale from 0-5 to describe a patient's level of functioning in terms of self care ability and activity level.
  0. Fully active
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature
  2. Ambulatory and capable of all self care but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited self care; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any self care; totally confined to bed or chair
  5. Dead
  Participants | 16

OUTCOME MEASURES:

1. Primary Outcome: Overall Tumor Response Rate as Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) Criteria. Sum of Partial Responses (PR) and Complete Responses (CR).
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions. Measurable lesions must be accurately measured in at least one dimension (longest diameter to be recorded) as > 20 mm with conventional techniques or as > 10mm with spiral CT scan or nonmeasurable, but evaluable. Evaluable is nonmeasurable disease that includes ascites, malignant pleural/pericardial effusion, bone lesions, or marrow involvement.
Time Frame: Baseline, after cycle 2, within 2 weeks of completing cycle 4
Measure: Count of Participants; unit: Participants
Arm/Group | Vinflunine + Cetuximab
Number analyzed (Participants) | 13
Participants | 3

2. Secondary Outcome: Duration of Response
Time Frame: After cycle 4
Population: Data not collected due to early study termination.
Arm/Group | Vinflunine + Cetuximab
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Survival
Time Frame: Every 30 days
Population: Data not collected due to early study termination.
Arm/Group | Vinflunine + Cetuximab
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression-free Survival
Time Frame: after cycle 2, within 2 weeks of completing cycle 4
Population: Data not collected due to early study termination.
Arm/Group | Vinflunine + Cetuximab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Patients were followed until disease progression, death, or six months after completion of treatment.
Arm/Group | Vinflunine + Cetuximab
All-Cause Mortality (participants affected / at risk) | 6/16
Serious Adverse Events (participants affected / at risk) | 8/16
Other Adverse Events (participants affected / at risk) | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vinflunine + Cetuximab (N=16)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 2
Infection - Lung (Infections and infestations) | 1 — Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L) - Lung (pneumonia)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 1
Thrombosis/embolism (vascular access-related) (Injury, poisoning and procedural complications) | 1
Constipation (Gastrointestinal disorders) | 2
Ileus, GI (functional obstruction of bowel, i.e., neuroconstipation) (Gastrointestinal disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vinflunine + Cetuximab (N=16)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Constipation (Gastrointestinal disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Creatinine (Investigations) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dry eye syndrome (Eye disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3
Fatigue (asthenia, lethargy, malaise) (General disorders) | 4
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 3
Hemorrhage, pulmonary/upper respiratory - Bronchopulmonary NOS (Respiratory, thoracic and mediastinal disorders) | 2
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 1
Hemorrhage, pulmonary/upper respiratory - Respiratory tract NOS (Respiratory, thoracic and mediastinal disorders) | 1
Leukocytes (total WBC) (Investigations) | 1
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 2
Metabolic/Laboratory - Other (Specify, __) (Metabolism and nutrition disorders) | 1 — Hyperbilirubinemia
Mood alteration - Anxiety (Psychiatric disorders) | 2
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 1
Nail changes (Skin and subcutaneous tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 11
Ocular/Visual - Other (Specify, __) (Eye disorders) | 2 — Red and tearing eye
Ophthalmoplegia/diplopia (double vision) (Eye disorders) | 1
Pain - Abdomen NOS (Gastrointestinal disorders) | 3
Pain - Chest/thorax NOS (General disorders) | 1
Pain - Other (Specify, __) (General disorders) | 1 — Joint/bone pain
Pain - Pain NOS (General disorders) | 5
Pain - Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 1
Pain - Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Platelets (Investigations) | 1
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1
Pulmonary/Upper Respiratory - Other (Specify, __) (Respiratory, thoracic and mediastinal disorders) | 1 — Chest congestion
Pulmonary/Upper Respiratory - Other (Specify, __) (Respiratory, thoracic and mediastinal disorders) | 1 — Hemoptysis
Rash/desquamation (Skin and subcutaneous tissue disorders) | 6
Rash: dermatitis associated with radiation - Chemoradiation (Injury, poisoning and procedural complications) | 1
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 1
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 1
Thrombosis/embolism (vascular access-related) (Injury, poisoning and procedural complications) | 1
Tremor (Nervous system disorders) | 1
Ulceration (Skin and subcutaneous tissue disorders) | 1
Vasovagal episode (Nervous system disorders) | 1
Vomiting (Gastrointestinal disorders) | 3

LIMITATIONS AND CAVEATS:
Study was terminated early due to unavailable drug/funding. Preliminary analysis reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days